CLINICAL TRIAL: NCT05908487
Title: African Americans (AA) Communities Speak: Partnering With AA in the North and South to Train Palliative Care Clinicians to Address Interpersonal and Systemic Racism and Provide Culturally Aligned Care.
Brief Title: African Americans (AA) Communities Speak
Acronym: AACS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Montefiore Medical Center (Other); University of California, San Francisco (Other); University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Ronit Elk, Associate Director, Center of Palliative and Supportive Care, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB300007677
Record Dates: First submitted 2023-06-01; First posted 2023-06-18 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Healthy Aging; Health Knowledge, Attitudes, Practice; Social Responsibility; Care Eliciting Behavior; Racism, Systemic
Keywords: goal concordant care older African American CBPR end-of-life
MeSH Terms: conditions — Behavior; Systemic Racism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Clinician Trainees- Cluster 1 (Other): Within each participating institution, clinician clusters are randomized to 1 of 4 start date training times for the African American Communities Speak (AACS) Education Intervention. Each arm has a pre-intervention (control) period and a post-intervention (exposure) period.
  Interventions: Behavioral: AA Communities Speak to Healthcare Professionals
- Clinician Trainees- Cluster 2 (Other): Within each participating institution, clinician clusters are randomized to 1 of 4 start date training times for the African American Communities Speak (AACS) Education Intervention. Each arm has a pre-intervention (control) period and a post-intervention (exposure) period
  Interventions: Behavioral: AA Communities Speak to Healthcare Professionals
- Clinician Trainees- Cluster 3 (Other): Within each participating institution, clinician clusters are randomized to 1 of 4 start date training times for the African American Communities Speak (AACS) Education Intervention. Each arm has a pre-intervention (control) period and a post-intervention (exposure) period
  Interventions: Behavioral: AA Communities Speak to Healthcare Professionals
- Clinician Trainees- Cluster 4 (Other): Within each participating institution, clinician clusters are randomized to 1 of 4 start date training times for the African American Communities Speak (AACS) Education Intervention. Each arm has a pre-intervention (control) period and a post-intervention (exposure) period
  Interventions: Behavioral: AA Communities Speak to Healthcare Professionals

INTERVENTIONS:
Behavioral: AA Communities Speak to Healthcare Professionals — The training program is designed to empower clinicians to improve goal-concordant EoL care delivery by using community-developed storytelling videos to create empathy with experiences of racism in EoL care, guidelines for culturally concordant EoL care delivery, and implicit bias recognition and management training to mitigate bias in goals of care communication.
  Other Names: Clinician Training

SUMMARY:
African Americans are less likely to receive quality end-of-life (EoL) care. Addressing disparities in EoL care will need efforts to support a better understanding of African American patients' EoL cultural values and preferences for EoL communication and the impact of historical and ongoing care delivery inequities in healthcare settings.

Our proposed "Caring for Older African Americans" training program is designed to empower clinicians to improve goal-concordant EoL care delivery by using community-developed storytelling videos to create empathy with experiences of racism in EoL care, guidelines for culturally concordant EoL care delivery, and an implicit bias recognition and management training to mitigate bias in goals of care communication.

DETAILED DESCRIPTION:
African Americans (AA) are less likely to receive quality end-of-life (EoL) care. For example, goals of care conversations, which are critical discussions between clinicians, patients, and families near the end of life, are less likely to occur for AAs than for Whites, and preferences are less likely to be followed when they do occur. Instead, families are more likely to be labeled as "difficult" if their decisions are incongruent with clinicians' recommendations. EoL decisions for many AA persons are rooted in both culture and a lifetime of experiences of structural racism. Efforts to address disparities need to address multiple factors such as patient-level cultural identity and EoL care values, interpersonal- and community-level norms for EoL communication and treatment, and healthcare institutional contexts for delivering EoL care in a setting affected by institutional racism.

Our research group began to address this need with 'African American Community Speaks', a proof-of-concept prototype of a community-developed training program for clinicians caring for AA older adults with serious illnesses. The program originally focused on rural Southern older AAs and is not broadly generalizable across the US due to geographic differences in culture, attitudes, and communication preferences among AA persons in the US. Thus, we propose to adapt our prototype program to urban-dwelling Southern and Northern older AA adults using our established platform of Community-Based Participatory Research (CBPR) in two geographically diverse regions: Birmingham, Alabama, and the Bronx, New York. To create the new training program called 'Caring for Older African Americans', our team of experts in CBPR, medical sociology, and clinical trials will work with local Community Advisory Boards to: 1. Conduct a comparative ethnographic study of urban dwelling AAs in the North and South to describe AA community values and preferences related to EoL care; 2. Adaptation of our prior community-developed training program by integrating community-developed storytelling videos for empathizing with experiences of racism in EoL care, guidelines for culturally concordant EoL care delivery, and adapting an existing implicit bias management program to goals of care communication; and 3. Conduct a cluster randomized trial in which we will randomize training times to 1 of 4 start dates using a stepped wedge design to accommodate the training of all clinicians and to mitigate the effect of secular trends.

Patients' personal experience of racism will be measured using the discrimination subscale of the Group Based Mistrust Scale. The primary outcome will be patient/family's perception of therapeutic alliance using The Human Connection Scale. Secondary outcomes will be family-reported goal-concordant care, and clinicians' knowledge of cultural values, awareness of implicit bias, and confidence to change practice. This innovative effort will be the first training program that: 1. addresses culturally concordant care, systemic racism, and implicit bias management, the three key elements in enhancing the provision of equitable care; and 2. is designed and implemented in full partnership with two distinct AA communities in the South and the North of the US.

ELIGIBILITY:
Inclusion Criteria: Aim 1.1

Person with serious Illness:

* Self-identified as African American (i.e., born, raised, and lived primarily in the US)
* Non-Hispanic or Latino
* Age ≥60 years
* English-speaking
* Has been diagnosed with a condition that fits into one of 3 illness paradigms including cancer, cardiac disease, pulmonary disease, neuro-degenerative disease, renal disease, stroke, sepsis, hepatic disease)
* Callahan Six-Item Screener score ≥4
* Able to complete baseline surveys.

Bereaved family member:

* Self-identified as African American (i.e., born, raised, and lived primarily in the US)
* Non-Hispanic or Latino
* Age ≥60 years
* English-speaking
* Loved one dies in the last 12 months and was diagnosed with a condition that fits into one of 3 illness paradigms including cancer, cardiac disease, pulmonary disease, neuro- degenerative disease, renal disease, stroke, sepsis, hepatic disease)
* Callahan Six-Item Screener score ≥4
* Able to complete baseline surveys.

Exclusion Criteria

Person with serious illness:

-Cannot be receiving hospice care

Bereaved Family Member:

-Cannot be a paid "sitter"

Inclusion Criteria: Aim 1.2

Bereaved Family member:

* Self-identified as African American (i.e., born, raised, and lived primarily in the US)
* Non-Hispanic or Latino
* Age ≥60 years
* English-speaking
* Loved one dies in the last 12 months and was diagnosed with a condition that fits into one of 3 illness paradigms including cancer, cardiac disease, pulmonary disease, neuro- degenerative disease, renal disease, stroke, sepsis, hepatic disease)
* Callahan Six-Item Screener score ≥4
* Able to complete baseline surveys

Pastors:

* Self-identifying as African American
* White, Non-Hispanic or Latino
* Sged ≥18 years old.

Inclusion Criteria: Aim 3

Clinician eligibility:

* Practice at a University of Alabama at Birmingham (UAB) or Montefiore/Einstein site that provides care to patients eligible for outcomes surveys
* At least 3 months of clinical practice at the study site prior to the intervention training to measure pre-intervention patient surveys

Exclusion criteria:

-Lack of at least 3 months of clinical practice at the study site prior to the intervention training.

Patient eligibility:

* Self-identified as African American (i.e., born, raised, and lived primarily in the US)
* Non-Hispanic or Latino, 3. age ≥60 years
* English-speaking
* Has been diagnosed with a condition that fits into one of 3 illness paradigms including cancer, cardiac disease, pulmonary disease, neuro-degenerative disease, renal disease, stroke, sepsis, hepatic disease)
* Callahan Six-Item Screener score ≥4
* Able to complete baseline surveys.

Exclusion criteria include:

-Currently receiving hospice care.

Family member eligibility:

* Age ≥ 18 years
* English-speaking
* Community-dwelling
* Unpaid care provider of a person with a serious illness.

Exclusion criteria: 1. Cannot be a paid "sitter".

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Human Connection Scale (patient/family reported) | up to 3 months before the intervention
  The Human Connection (THC) Scale is a summary score of item responses such that a higher total score indicates greater therapeutic alliance. Possible scores range from 16 to 64. The 16-item THC scale had a high degree of internal consistency (Cronbach α= 90).
Human Connection Scale (patient/ family reported) | up to 3 months after intervention
  The Human Connection (THC) Scale is a summary score of item responses such that a higher total score indicates greater therapeutic alliance. Possible scores range from 16 to 64. The 16-item THC scale had a high degree of internal consistency (Cronbach α= 90).

SECONDARY OUTCOMES:
Goal Concordant Care (patient/family reported) | up to 3 months before the intervention
  Goal Concordant Care will be measured based on responses to the following two questions, each with a dichotomous outcome: 1. Family member reports that the patient's end-of-life wishes were adequately discussed with the family respondent 2. Family member's satisfaction that patient's end-of-life were met.
  Johnson, S.B., Butow, P.N., Bell, M.L. et al. A randomized controlled trial of an advance care planning intervention for patients with incurable cancer. Br J Cancer 119, 1182-1190 (2018).
  https://doi.org.10.1038/s41416-018-0303-7
Goal Concordant Care (patient/family reported) | up to 3 months after the intervention
  Goal Concordant Care will be measured based on responses to the following two questions, each with a dichotomous outcome: 1. Family member reports that the patient's end-of-life wishes were adequately discussed with the family respondent 2. Family member's satisfaction that patient's end-of-life were met.
  Johnson, S.B., Butow, P.N., Bell, M.L. et al. A randomized controlled trial of an advance care planning intervention for patients with incurable cancer. Br J Cancer 119, 1182-1190 (2018).
  https://doi.org.10.1038/s41416-018-0303-7

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Tjia, MD, MSCE, Principal Investigator — University of Massachusetts, Worcester
Locations (3):
- United States (3):
  - UAB, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Albert Einstein/Montefiore, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No